CLINICAL TRIAL: NCT04557644
Title: Contagious Itch, Disgust and Empathy in Patients and Medical Staff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: sp20Mueller; 2020-01089
Record Dates: First submitted 2020-09-15; First posted 2020-09-21 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Contagious Itch
Keywords: itch; scabies; ectoparasites; post-scabetic itch; disgust; empathy
MeSH Terms: conditions — Pruritus; Scabies | interventions — Functional Status

STUDY DESIGN:
Intervention Model Description: In this study both the staff and the infested family are to complete questionnaires addressing CI, disgust and empathy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- medical staff treating patients with scabies (Active Comparator)
  Interventions: Other: 7-items-questionnaires addressing CI, disgust and empathy; Other: Saarbrucken Personality questionnaire (SPQ) addressing empathy.
- family infested with scabies (Active Comparator)
  Interventions: Other: Saarbrucken Personality questionnaire (SPQ) addressing empathy.; Other: 10-items-questionnaire addressing previous dermatological conditions, intensity of itch; Other: ItchyQol-questionnaire composed of 22 items addressing itch-related symptoms, functions and emotions

INTERVENTIONS:
Other: 7-items-questionnaires addressing CI, disgust and empathy — 7-items-questionnaire including numerical rating scales (NRS) ranging from 0 (no itch/disgust/empathy) to 10 (worst itch/disgust/most empathy imaginable) to rate itch, disgust and empathy they experience when treating the infested families.
  Arms: medical staff treating patients with scabies
Other: Saarbrucken Personality questionnaire (SPQ) addressing empathy. — Empathy is additionally assessed by the Saarbrucken Personality Questionnaire (SPQ) ,a 16-item tool.
Other: 10-items-questionnaire addressing previous dermatological conditions, intensity of itch — 10-items-questionnaire (completed by the hospitalised family) regarding demographic information (gender, age, profession), previous dermatological conditions, intensity of itch a.) on the first day of the hospitalisation, b.) when seeing the skin lesions of the other family members c.) when talking about the scabies/itch with the other family members, d.) when seeing other family members scratching themselves, and questions regarding their intensity of disgust of the scabies and empathy for the other family members (0-10 NRS).
  Arms: family infested with scabies
Other: ItchyQol-questionnaire composed of 22 items addressing itch-related symptoms, functions and emotions — ItchyQol-questionnaire to assess the itch-related quality of life impairment. The ItchyQoL is composed of 22 items addressing itch-related symptoms, functions and emotions.
  Arms: family infested with scabies

SUMMARY:
This study is to assess the relationship between CI, disgust and empathy in medical staff treating patients with scabies, to differentiate the impact of visual and verbal stimuli contributing to CI and to assess information about CI, disgust and empathy in a family infested with scabies.

DETAILED DESCRIPTION:
Itch is the commonest skin-related symptom, defined as a bodily sensation provoking the urge to scratch. The induction of itch and scratching by mere (audio-) visual stimuli such as pictures of insects on skin or video clips showing individuals scratching themselves, indicates that itch can be perceived in the absence of a pruritogenic somatosensory stimulus. This phenomenon is referred to as "contagious itch" (CI). CI may play a special role in the content of scabies both for the affected patients as well as the treating staff: It is a very common phenomenon that family members who are not infested by scabies themselves experience itch when watching their infested relatives scratching. The same is very frequently expressed by health care professionals being confronted with scabies patients. Two further important factors may be involved in the context of CI: disgust and empathy. Empathy is defined as a psychological concept that enables individuals to understand and share emotions of others. Disgust is an emotional response of revulsion to potentially contagious and/or harmful objects or subjects. This study is to assess the relationship between CI, disgust and empathy in medical staff treating patients with scabies, to differentiate the impact of visual and verbal stimuli contributing to CI and to assess information about CI, disgust and empathy in a family infested with scabies.

ELIGIBILITY:
Inclusion Criteria:

* members of families (aged >7 years) hospitalized in the Department of Dermatology with scabies
* staff (physicians, nurses, nurse aids aged >16 years) involved in the treatment of these families
* Infestation of scabies in individual family members confirmed by two leading dermatologists of the University Hospital Basel by dermoscopy and/or skin scrapings.

Exclusion Criteria:

-

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Intensity of emotion (CI, disgust and empathy) in medical staff treating patients with scabies | one point assessment at baseline
  Score in 7-items-questionnaire including numerical rating scales (NRS) ranging from 0 (no itch/disgust/empathy) to 10 (worst itch/disgust/most empathy imaginable) to rate itch, disgust and empathy they experience when treating the infested families. The questionnaire (see Appendix) contains questions regarding demographic information (gender, age, profession), previous dermatological conditions, intensity of itch a.) before interacting with the patients, b.) when listening to the patients telling about their infestation with scabies, c.) when seeing the skin lesions, d.) when seeing patients scratching themselves, and questions regarding their intensity of disgust of the scabies and empathy for the families (0-10 NRS).
Intensity of emotion (CI, disgust and empathy) in family infested with scabies | one point assessment at baseline (first day of hospitalisation)
  Score in 10-items-questionnaire addressing intensity of itch a.) on the first day of their hospitalisation, b.) when seeing the skin lesions of the other family members c.) when talking about the scabies/itch with the other family members, d.) when seeing other family members scratching themselves and intensity of disgust of the scabies and intensity of empathy for the other family members (0-10 NRS).
Empathy scored by Saarbrucken Personality Questionnaire (SPQ) | one point assessment at baseline (first day of hospitalisation)
  The Saarbrucken personality questionnaire SPQ is the German version of the Interpersonality Reactivity Index (IRI) used for the measurement of empathy. The tool is a self-report answered on a 5-point Likert scale ranging from "Does not describe me well" to "Describes me very well".

CONTACTS AND LOCATIONS:
Overall Officials: Simon Mueller, PD Dr. med., Principal Investigator — Department of Dermatology, University Hospital Basel
Locations (1):
- Department of Dermatology; University Hospital Basel, Basel, Switzerland